CLINICAL TRIAL: NCT07235813
Title: Estimation of Serum and Tissue Level of Interleukin-35 (IL-35) in Mycosis Fungoides Before and After Treatment
Brief Title: IL-35: A Key Immunosuppressive Driver in Mycosis Fungoides Modulated by Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, heba ahmed abdelgayed ibrahim, Lecturer of Dermatology, Cairo University, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-384-2024
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phototherapy Arm (Mycosis Fungoides Patients) (Experimental): Phototherapy Arm (Mycosis Fungoides Patients)
  Interventions: Radiation: Phototherapy (PUVA or NB-UVB)

INTERVENTIONS:
Radiation: Phototherapy (PUVA or NB-UVB) — Patients with mycosis fungoides will receive phototherapy three times per week. Most will undergo psoralen plus UVA (PUVA) with dose escalation based on skin phototype and tolerance. A minority may receive narrowband UVB (NB-UVB) following standard protocols. Treatment continues until lesion resolution or a maximum of 36 sessions. Blood and skin samples are collected before and after treatment to measure IL-35 levels.

SUMMARY:
Mycosis fungoides is the most common type of skin lymphoma. It develops when certain white blood cells (T cells) grow abnormally in the skin, causing red, scaly, or itchy patches. The disease is often treated with phototherapy, a light-based treatment that can control symptoms in early stages.

This study looked at a protein called interleukin-35 (IL-35), which normally helps regulate the immune system but can also suppress the body's ability to fight cancer. The investigators aimed to determine if IL-35 levels are higher in patients with mycosis fungoides and whether phototherapy can change those levels.

The study enrolled 16 patients with mycosis fungoides and compared them to 16 healthy people. Blood samples and small skin biopsies were taken before and after phototherapy. The study found that IL-35 levels were significantly higher in patients than in healthy people. After phototherapy, IL-35 levels dropped back to normal.

These results suggest that phototherapy not only treats skin lesions directly but also helps restore immune balance by lowering IL-35. IL-35 may become a useful marker to monitor disease activity and treatment response in patients with mycosis fungoides.

DETAILED DESCRIPTION:
Mycosis fungoides (MF) is the most common primary cutaneous T-cell lymphoma and is characterized by progressive immune dysregulation. Early disease often shows a T helper 1 (Th1) profile, while advanced stages shift toward an immunosuppressive T helper 2 (Th2) environment that promotes tumor persistence. Interleukin-35 (IL-35), a recently described member of the IL-12 cytokine family, has emerged as a potent immunosuppressive cytokine. It contributes to tumor growth by suppressing anti-tumor T-cell responses, expanding regulatory T cells, and fostering angiogenesis. Elevated IL-35 levels have been reported in several malignancies, including MF, but its behavior under therapeutic intervention has not been well defined.

Phototherapy, including psoralen plus ultraviolet A (PUVA) and narrowband ultraviolet B (NB-UVB), remains a cornerstone treatment for early-stage MF. Beyond its direct cytotoxic effects on malignant T cells, phototherapy exerts broad immunomodulatory actions on the cutaneous cytokine milieu. Prior studies have shown normalization of cytokines such as IL-15 following phototherapy, suggesting that its benefits extend beyond lesion clearance to restoration of immune balance.

This prospective interventional cohort study was designed to evaluate whether IL-35 levels in serum and skin tissue are altered by phototherapy in MF patients. Sixteen patients with histologically confirmed MF and sixteen matched healthy controls were enrolled. IL-35 was measured at baseline in both groups and again after phototherapy in patients. The study demonstrated that IL-35 levels were significantly elevated in MF patients compared to controls, and that both serum and tissue IL-35 declined after phototherapy, normalizing to control levels. These findings suggest that phototherapy may correct the immunosuppressive environment characteristic of MF, and that IL-35 could serve as a biomarker for disease activity and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mycosis fungoides; newly diagnosed or recurrent after cessation of treatment
* Both genders
* Age group ≥ 18 years old

Exclusion Criteria:

* Patients with any contraindication to phototherapy (e.g., any other skin cancers or photosensitivity); or to psoralen (e.g., liver disease).
* Subjects with history of solid or hematological malignancy as leukemia.
* Patients with autoimmune disease as SLE.
* Patients who received treatment for the past one month.
* Pregnant and lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in serum and tissue interleukin-35 (IL-35) levels in mycosis fungoides patients before and after phototherapy | Baseline and after up to 36 phototherapy sessions (approximately 3 months)
  Serum IL-35 concentration (ng/ml) measured by ELISA and tissue IL-35 concentration (ng/g) measured from skin biopsy homogenates. Samples collected at baseline and after completion of phototherapy (PUVA or NB-UVB). The primary endpoint is the difference in IL-35 levels pre- and post-treatment.

SECONDARY OUTCOMES:
Correlation between IL-35 levels and patient age | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between IL-35 levels (serum and tissue, baseline and post-treatment) and patient age in mycosis fungoides patients using Pearson or Spearman correlation analysis.
Correlation between IL-35 levels and disease extent | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between IL-35 levels (serum and tissue, baseline and post-treatment) and disease extent (measured by body surface area percentage) in mycosis fungoides patients using Pearson or Spearman correlation analysis.
Correlation between serum and tissue IL-35 levels | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between serum IL-35 concentration (ng/ml) and tissue IL-35 concentration (ng/g) at baseline and following phototherapy in mycosis fungoides patients using Pearson or Spearman correlation analysis.
Correlation between IL-35 levels and lactate dehydrogenase (LDH) | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between IL-35 levels (serum and tissue, baseline and post-treatment) and serum lactate dehydrogenase levels in mycosis fungoides patients using Pearson or Spearman correlation analysis.
Correlation between IL-35 levels and beta-2 microglobulin | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between IL-35 levels (serum and tissue, baseline and post-treatment) and serum beta-2 microglobulin levels in mycosis fungoides patients using Pearson or Spearman correlation analysis.
Correlation between IL-35 levels and disease duration | Baseline and after completion of phototherapy (up to 36 sessions, approximately 3 months)
  Assessment of the relationship between IL-35 levels (serum and tissue, baseline and post-treatment) and disease duration in mycosis fungoides patients using Pearson or Spearman correlation analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, English (English), Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center study with a small sample size, and de-identification cannot be fully guaranteed. Aggregate results, including summary statistics and outcome analyses, will be made available through publication